CLINICAL TRIAL: NCT05935774
Title: Phase 2 Trial of TGF-β2 Inhibition (OT-101) With Atezolizumab as Second-Line or Third-Line Therapy for Patients Previously Treated With Immunotherapy (+/- Chemotherapy) With Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: OT-101 in Combination With Atezolizumab for the Treatment of Metastatic or Recurrent Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn prior to opening to accrual.
Sponsor: University of Washington (Other)
Collaborators: Genentech, Inc. (Industry); Oncotelic Therapeutics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1123580; NCI-2023-04564 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1123580 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Biopsy; Magnetic Resonance Spectroscopy; Trabedersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (atezolizumab, trabedersen) (Experimental): Patients recieve atezolizumab IV on day 1 and trabedersen continuous IV on days 1-4 and days 15-19 of each cycle. Cycles repeat every 28 days for 104 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI during screening and every 8 weeks for the first 24 weeks and then every 12 weeks thereafter. Patients undergo blood sample collection prior to initiation of therapy, on day 4 of cycles 1-4, prior to weeks 4 and 8 of therapy, and at time of progression. Patients may also undergo biopsy during screening and/or 6-8 weeks after initiation of therapy.
  Interventions: Biological: Atezolizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Electronic Health Record Review; Procedure: Magnetic Resonance Imaging; Drug: Trabedersen (OT-101)

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL328OA; RG7446; RO5541267; Tecentriq
Procedure: Biopsy — Undergo biopsy
  Other Names: Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure)
Other: Electronic Health Record Review — Ancillary studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Trabedersen (OT-101) — Given IV
  Other Names: AP 12009

SUMMARY:
This phase II trial tests how well trabedersen (OT-101) in combination with atezolizumab works in treating patients with non-small cell lung cancer (NSCLC) that has spread from where it first started (lung) to other places in the body (metastatic) or has come back after a period of improvement (recurrent). OT-101 is a transforming growth factor (TGF)-beta2 specific drug. TGF-beta2, a cytokine that is often overexpressed in various malignant tumors, may play an important role in promoting the growth, progression and migration of tumor cells. OT-101 binds to the TGF-beta2 receptor causing inhibition of protein production, thereby decreasing TGF-beta2 protein levels which may result in the inhibition of tumor cell growth and migration. Atezolizumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Giving OT-101 and atezolizumab together may be an effective treatment for patients with metastatic or recurrent NSCLC.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive atezolizumab intravenously (IV) on day 1 and trabedersen continuous IV on days 1-4 and days 15-19 of each cycle. Cycles repeat every 28 days for 104 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and every 8 weeks for the first 24 weeks and then every 12 weeks thereafter. Patients undergo blood sample collection prior to initiation of therapy, on day 4 of cycles 1-4, prior to weeks 4 and 8 of therapy, and at time of progression. Patients may also undergo biopsy during screening and/or 6-8 weeks after initiation of therapy.

After completion of study treatment, patients are followed up to 90 days and then every 3 months for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and older
* Pathologically or cytologically confirmed non-small cell lung cancer with no known targetable genomic alterations with Food and Drug Administration (FDA) approved targeted therapies: including EGFR mutation, ALK rearrangement, ROS1 rearrangements MET or RET fusions, BRAF mutations, HER2 mutations or NTRK fusion
* Metastatic or recurrent NSCLC who have received prior immune checkpoint inhibitor and chemotherapy (in first or second line) for metastatic or recurrent disease and have had at least one prior line of cancer directed therapy

  * Minimum duration on first-line immune checkpoint inhibitor (ICI) is 84 days (cannot have had progressive disease [PD] as best response)
* At least one site of measurable disease as determined by the Investigator, using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria. Participants must have measurable disease, defined as at least one lesion that can be measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1. Participants must have ECOG PS 0 or 1 at the time of informed consent and at the time of treatment initiation

  * NOTE: Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention
* Must be willing to provide pre-treatment archived specimen or undergo a biopsy procedure if archived specimen is not available or if > 6 months old
* Must be willing to provide an on-treatment biopsy, if deemed safe by the treating physician. If deemed unsafe by the treating physician, the on-treatment biopsy requirement will be waived
* Platelet count >= 100,000/uL
* Absolute neutrophil count >= 1,500/uL
* Hemoglobin >= 9g/dL (transfusions are allowed if done before 14 days of measurement)
* Serum albumin >= 25 g/L (2.5 g/dL)
* For patients not receiving therapeutic anticoagulation: International normalized ratio (INR) or activated partial thromboplastin time (aPTT) =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times upper limit of normal, in the presence of liver metastasis AST and ALT =< 5 times upper limit of normal
* Total bilirubin =< 1.5 x ULN; no history of Gilberts disease
* Creatinine clearance (CrCl) > 60 mL/min
* Baseline electrocardiography (ECG) with corrected QTc < 480 msec (using QTcF or Fridericia correction formula for QTC which can be found on MD Calc)
* Women of child-bearing potential and sexually active men must agree to use adequate contraception (hormonal or barrier method) prior to treatment initiation, during treatment and for three months after completing treatment
* Negative beta-human chorionic gonadotropin (hCG) pregnancy test at screening for women of childbearing potential. Pregnant or breast feeding women are not eligible
* Ability to understand and willingness to sign a written and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrollment
* For patients receiving therapeutic anticoagulation: Stable anticoagulant regimen
* Negative human immunodeficiency virus (HIV) test at screening, with the following exception: Patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count >= 200/uL, and have an undetectable viral load
* Negative hepatitis B screening as below:

  * Negative hepatitis B surface antigen (HBsAg) test at screening
  * Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) deoxyribonucleic acid (DNA) test at screening
  * The HBV DNA test will be performed only for patients who have a negative hepatitis B virus surface antigen (HBsAg) test and a positive total HBcAb test
* Negative Hepatitis C screening as below:

  * Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV ribonucleic acid (RNA) test at screening
  * The HCV RNA test must be performed for patients who have a positive HCV antibody test

Exclusion Criteria:

* Participants who have had chemotherapy or systemic therapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. NOTE: Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy are eligible. Participants with endocrine-related AEs grade =< 2 requiring treatment or hormone replacement are eligible
* Patients for whom best response to 1 line (L ) or 2L treatment with was progressive disease within 84 days of treatment
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities and not have had radiation pneumonitis
* Surgery within 21 days of start of study treatment. Minor surgery within 2 weeks of start of study treatment. Placement of vascular access device and biopsies are not considered major or minor surgery and are allowed
* Has a history of a second invasive malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. All patients with previously treated in situ carcinoma are eligible, as patients with history of non-melanoma skin cancer
* Symptomatic central nervous system (CNS) metastases; participants with known brain metastasis must be asymptomatic with no steroids or antiepileptics within 7 days prior to start of study treatment

  * Patients with untreated CNS metastases may be enrolled as long as they meet the above criteria. Patients with bulky CNS metastases should consider receiving radiation prior to study entry per investigator judgment
* Participants with spinal cord compression must have received local treatment and must have been symptomatically stable with no use of steroids for at least 7 days prior to start of study treatment
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
  * Participants must not have an active autoimmune disease that has required immune modulating treatment within two years prior to consenting (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs)
  * Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed
* Known history of primary immunodeficiency
* History of allogeneic tissue/solid organ transplant that requires use of immunosuppressives
* Current symptomatic pneumonitis and any past history of immune checkpoint inhibitor related pneumonitis regardless of steroid treatment history
* Severe lung disease (e.g., chronic obstructive pulmonary disease [COPD] or interstitial lung disease [ILD]) who cannot stop steroids 7 days prior to start of study treatment
* Serious cerebrovascular and cardiac disease (such as New York Heart Association class II or greater cardiac disease) defined as:

  * Active unstable angina pectoris
  * Congestive heart failure NYHA (New York Heart Association) > grade 3
  * Acute myocardial infarction within 3 months of consenting
  * Stroke or transient ischemic attack within 3 months of consenting
* Known active chronic infections: Active hepatitis B, hepatitis C and tuberculosis. Active infection requiring IV antibiotics within 7 days of study treatment initiation
* Uncontrolled or concurrent illness, laboratory abnormality, psychiatric illness/social situations, or any condition that would limit compliance with study requirements or is not in the best interest of the participant to participate in the opinion of the treating investigator
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 150 days after the last dose of trial treatment
* Prior allergic reactions or severe hypersensitivity (>= grade 3) to compounds similar to the investigational agents
* History of leptomeningeal disease
* Uncontrolled tumor-related pain

  * Patients requiring pain medication must be on a stable regimen at study entry
  * Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period
  * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

  * Patients with indwelling catheters (e.g., PleurX [registered trademark]) are allowed
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Treatment with investigational therapy within 28 days prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 60 months
  Objective response measured by Response Evaluation Criteria in Solid Tumors version 1.1 defined as a confirmed or unconfirmed complete or partial response. Continuous outcomes will be summarized descriptively by means, medians, and quantiles. For the primary analyses, binary proportions will be estimated along with 90% confidence intervals.

SECONDARY OUTCOMES:
Duration of response | From first documented response to progressive disease, symptomatic deterioration, or death due to any cause in responder subset, assessed up to 60 months
  Distributions of time-to-event outcomes will be estimated using Kaplan-Meier. Confidence intervals about medians will be estimated using the Brookmeyer-Crowley method.
Disease control rate | At 6 months from treatment initiation
  Measured by complete response, partial response, and stable disease. Continuous outcomes will be summarized descriptively by means, medians, and quantiles. For the primary analyses, binary proportions will be estimated along with 90% confidence intervals.
Progression free survival | Duration between treatment initiation and progressive disease, symptomatic deterioration, or death due to any cause, whichever occurs first, assessed up to 60 months
  Distributions of time-to-event outcomes will be estimated using Kaplan-Meier. Confidence intervals about medians will be estimated using the Brookmeyer-Crowley method.
Overall survival | From the date of treatment initiation to date of death due to any cause, assessed up to 60 months
  Distributions of time-to-event outcomes will be estimated using Kaplan-Meier. Confidence intervals about medians will be estimated using the Brookmeyer-Crowley method.
Incidence of adverse events | Up to 90 days
  Safety defined at toxicity grade and attribution by Common Terminology Criteria for Adverse Events 5.0. Continuous outcomes will be summarized descriptively by means, medians, and quantiles. For the primary analyses, binary proportions will be estimated along with 90% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Santana-Davila, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No